CLINICAL TRIAL: NCT02124148
Title: A Phase 1b Trial of LY2606368 in Combination With Chemotherapy or Targeted Agents in Advanced and/or Metastatic Tumors
Brief Title: A Study of Prexasertib (LY2606368) With Chemotherapy or Targeted Agents in Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15295; I4D-MC-JTJF (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Neoplasm Metastasis; Colorectal Neoplasms; Breast Cancer
Keywords: cancer
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Breast Neoplasms; Neoplasms | interventions — prexasertib; Cisplatin; Cetuximab; Granulocyte Colony-Stimulating Factor; Pemetrexed; Fluorouracil; LY3023414; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Prexasertib + Cisplatin (Part A) (Experimental): Part A: Prexasertib and cisplatin administered intravenously (IV) once every 21 days.
  Part A2: Prexasertib and cisplatin administered IV every 21 days; G-CSF administered subcutaneously (SC) starting approximately 24 hours after each prexasertib dose every 21 days.
  Part A3: Cisplatin administered IV on day one and prexasertib administered IV on day two once every 21 days.
  Part A Expansion: Part A, A2, and/or A3 may be expanded at the recommended dose.
  Participants may remain on treatment until discontinuation criteria are met.
  Interventions: Drug: Prexasertib; Drug: Cisplatin; Drug: G-CSF
- Prexasertib + Cetuximab (Part B) (Experimental): Part B: Cetuximab administered IV weekly and prexasertib administered IV once every 14 days.
  Part B2: Cetuximab administered IV weekly and prexasertib administered IV once every 14 days; G-CSF administered SC starting approximately 24 hours after each prexasertib dose every 14 days.
  Part B3: Cetuximab administered IV with prexasertib administered IV once every 14 days.
  Part B Expansion: Part B, B2 and/or B3 may be expanded at the recommended dose.
  Participants may remain on treatment until discontinuation criteria are met.
  Interventions: Drug: Prexasertib; Drug: Cetuximab; Drug: G-CSF
- Prexasertib + Pemetrexed (Part C) (Experimental): Part C: Pemetrexed administered IV on day one and prexasertib administered IV on day one and two every 21 days.
  Participants may remain on treatment until discontinuation criteria are met.
  Interventions: Drug: Prexasertib; Drug: Pemetrexed
- Prexasertib + 5-FU (Part D) (Experimental): Part D: Leucovorin administered IV on day one, 5-FU administered IV bolus on day one and by continuous IV on days one to three (46 hours), and prexasertib administered IV on day three every 14 days.
  Participants may remain on treatment until discontinuation criteria are met.
  Interventions: Drug: Prexasertib; Drug: Fluorouracil; Drug: Leucovorin
- Prexasertib + LY3023414 (Part E) (Experimental): Part E: Prexasertib administered IV on day one and LY3023414 administered orally twice daily every 14 days.
  Part E will be expanded at the recommended dose in participants with advanced or metastatic cancer, participants with PIK3CA mutations (E2 expansion), or with advanced or metastatic ER-negative, PR-negative, and HER-2 non-overexpressing breast cancer (E3 expansion).
  Participants may remain on treatment until discontinuation criteria are met.
  Interventions: Drug: Prexasertib; Drug: LY3023414

INTERVENTIONS:
Drug: Prexasertib — Administered IV
  Other Names: LY2606368
Drug: Cisplatin — Administered IV
  Arms: Prexasertib + Cisplatin (Part A)
Drug: Cetuximab — Administered IV
  Other Names: Erbitux
  Arms: Prexasertib + Cetuximab (Part B)
Drug: G-CSF — Administered SC
  Arms: Prexasertib + Cetuximab (Part B); Prexasertib + Cisplatin (Part A)
Drug: Pemetrexed — Administered IV
  Other Names: Alimta
  Arms: Prexasertib + Pemetrexed (Part C)
Drug: Fluorouracil — Administered IV
  Arms: Prexasertib + 5-FU (Part D)
Drug: LY3023414 — Administered PO
  Arms: Prexasertib + LY3023414 (Part E)
Drug: Leucovorin — Administered IV
  Arms: Prexasertib + 5-FU (Part D)

SUMMARY:
The main purpose of this study is to investigate the safety of prexasertib in combination with other anti-cancer drugs (cisplatin, cetuximab, pemetrexed, fluorouracil or LY3023414) in participants with advanced cancer or cancer that has spread to another part of the body. The study has multiple parts (A, B, C, D and E). Participants will only enroll in one part.

DETAILED DESCRIPTION:
The primary purpose of Parts A, B, C, D and E of this study is to determine a recommended dose level and schedule of prexasertib (an inhibitor of checkpoint kinase 1 and 2 [CHK1/CHK2] in combination with:

* cisplatin (Part A)
* cetuximab (Part B)
* pemetrexed (Part C)
* fluorouracil (Part D)
* LY3023414 (Part E) [An inhibitor of phosphoinositide 3-kinase alpha (PI3K alpha) and mammalian target of rapamycin (mTOR), DNA-dependent protein kinase (DNA-PK), and other class I phosphoinositide 3-kinase (PI3K) family members]

in participants with advanced or metastatic cancer.

Part A dose expansion of the study will evaluate the safety and toxicity of prexasertib at the recommended dose level in combination with cisplatin in participants with advanced or metastatic cancer, Part B dose expansion of the study will evaluate the safety and toxicity of prexasertib at the recommended dose level in combination with cetuximab in participants with advanced or metastatic colorectal cancer, Part C and D dose expansions have been removed and Part E dose expansion of the study will evaluate the safety and toxicity of prexasertib at the recommended dose level in combination with LY3023414 in participants with advanced or metastatic cancer, participants with PIK3CA mutations, or with advanced or metastatic breast cancer.

In Parts A and B the effect of adding granulocyte colony stimulating factor (G-CSF) to cisplatin in combination with prexasertib and cetuximab in combination with prexasertib will be explored. In Part A the effect of changing the schedule of prexasertib and cisplatin also will be explored. In Part B the effect of changing the schedule of prexasertib and cetuximab also will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Must be appropriate candidate for experimental therapy, as determined by investigator, after available standard therapies have failed
* Have adequate organ function
* Prior Therapies: Systemic treatments: must have discontinued previous systemic treatments for cancer and recovered from the acute effects of therapy. Participants must have discontinued mitomycin-C or nitrosourea therapy at least 42 days and have discontinued any cytotoxic therapies at least 28 days prior to study enrollment. Radiation therapy and surgery: must be completed at least 4 weeks before study enrollment
* All parts except Part B, Part E2, and Part E3 dose expansion: Must have diagnosis of cancer that is advanced or metastatic
* Part B dose expansion: Must have confirmed Kirsten rat sarcoma viral oncogene homolog (KRAS) wild-type colorectal cancer that is metastatic or recurrent and has failed oxaliplatin- and irinotecan-based chemotherapy or who are intolerant of irinotecan or oxaliplatin
* Part E2 dose expansion: must have cancer that is advanced or metastatic and have prior documentation of a mutation of PIK3CA
* Part E3 dose expansion: must have advanced or metastatic ER-negative, PR-negative, and HER-2 non-overexpressing breast cancer
* Must be available during the duration of the study and willing to follow the study procedures
* Parts A and B: If participant is of reproductive potential, must agree to use medically approved contraceptive precautions during the study and for six months following the last dose of study drug
* Parts C, D and E: If participant is of reproductive potential, must agree to use medically approved contraceptive precautions during the study and for three months following the last dose of study drug
* If the participant is a female of childbearing potential, must have had a negative serum or urine pregnancy test within 14 days of the first dose of study drug and must not be breast feeding
* Part E: Are able to swallow capsules or tablets

Exclusion Criteria:

* Have received more than 2 previous lines of cytotoxic chemotherapy (if receiving cisplatin, 5-FU or pemetrexed)
* Must not have taken an unapproved drug as treatment for any indication within the last 28 days prior to starting study treatment
* Must not have an active symptomatic fungal, bacterial or viral infection, including human immunodeficiency virus (HIV) or Hepatitis A, B, or C
* Must not have a serious heart condition, such as congestive heart failure, unstable angina pectoris, or heart attack within the last three months
* Must not have a family history of long QTc syndrome
* Must not have a serotonin-secreting carcinoid tumor or a prior history of drug-induced serotonin syndrome
* Must not have acute leukemia
* Part E: Have insulin-dependent (type I) diabetes or a history of gestational diabetes
* Part E: Prior treatment with a PI3K/mTOR inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2014-06-18 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Tolerated Dose and Schedule of Prexasertib in Combination with Cisplatin | Cycle 1 predose through last dose last cycle (estimated up to 24 weeks)
Part B: Maximum Tolerated Dose of Prexasertib in Combination with Cetuximab | Cycle 1 predose through last dose last cycle (estimated up to 24 weeks)
Part C: Maximum Tolerated Dose of Prexasertib in Combination with Pemetrexed | Cycle 1 predose through last dose last cycle (estimated up to 24 weeks)
Part D: Maximum Tolerated Dose of Prexasertib in Combination with Fluorouracil (5-FU) | Cycle 1 predose through last dose last cycle (estimated up to 24 weeks)
Part E: Maximum Tolerated Dose of Prexasertib in Combination with LY3023414 | Cycle 1 predose through last dose last cycle (estimated up to 24 weeks)

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Plasma Concentration of Prexasertib | Cycle 1 Predose through Cycle 2, Day 15
Pharmacokinetics: Area Under the Plasma Concentration Curve of Prexasertib | Cycle 1 Predose through Cycle 2, Day 15
Pharmacokinetics: Maximum Plasma Concentration of Cisplatin (Total Platinum) | Cycle 1 Predose through Cycle 2, Day 1
Pharmacokinetics: Area Under the Plasma Concentration Curve of Cisplatin (Total Platinum) | Cycle 1 Predose through Cycle 2, Day 1
Pharmacokinetics: Maximum Plasma Concentration of Cetuximab | Cycle 1 Predose through Cycle 3, Day 1
Pharmacokinetics: Maximum Plasma Concentration of Pemetrexed | Cycle 1 Predose through Cycle 1, Day 2
Pharmacokinetics: Area Under the Plasma Concentration Curve of Pemetrexed | Cycle 1 Predose through Cycle 1, Day 2
Pharmacokinetics: Maximum Plasma Concentration of 5-FU | Cycle 1 Predose through Cycle 1, Day 3
Pharmacokinetics: Maximum Plasma Concentration of LY3023414 | Cycle 1 Predose through Cycle 2, Day 2
Pharmacokinetics: Area Under the Plasma Concentration Curve of LY3023414 | Time Frame: Cycle 1 Predose through Cycle 2, Day 2
B2, E2, E3 Dose Expansion: Overall Response Rate | Baseline through disease progression (estimated as up to 24 weeks) or death from any cause
B2, E2, E3 Dose Expansion: Disease Control Rate | Baseline through disease progression (estimated as up to 24 weeks) or death from any cause
B2, E2, E3 Dose Expansion: Progression-Free Survival | Baseline through disease progression (estimated as up to 24 weeks) or death from any cause
B2, E2, E3 Dose Expansion: Duration of Response | Baseline through disease progression (estimated as up to 24 weeks) or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Florida Cancer Specialists, Sarasota, Florida
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute SCRI, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Moore KN, Hong DS, Patel MR, Pant S, Ulahannan SV, Jones S, Meric-Bernstam F, Wang JS, Aljumaily R, Hamilton EP, Wittchen ES, Wang X, Lin AB, Bendell JC. A Phase 1b Trial of Prexasertib in Combination with Standard-of-Care Agents in Advanced or Metastatic Cancer. Target Oncol. 2021 Sep;16(5):569-589. doi: 10.1007/s11523-021-00835-0. Epub 2021 Sep 24. PMID 34559360
- [Derived] Hong DS, Moore KN, Bendell JC, Karp DD, Wang JS, Ulahannan SV, Jones S, Wu W, Donoho GP, Ding Y, Capen A, Wang X, Bence Lin A, Patel MR. Preclinical Evaluation and Phase Ib Study of Prexasertib, a CHK1 Inhibitor, and Samotolisib (LY3023414), a Dual PI3K/mTOR Inhibitor. Clin Cancer Res. 2021 Apr 1;27(7):1864-1874. doi: 10.1158/1078-0432.CCR-20-3242. Epub 2021 Jan 25. PMID 33495309
- See also: A Study of Prexasertib (LY2606368) With Chemotherapy or Targeted Agents in Participants With Advanced Cancer — https://www.lillytrialguide.com/en-US/studies/solid-tumor/JTJF#?postal=